CLINICAL TRIAL: NCT04050046
Title: Noninvasive Brain Stimulation to Enhance Cognitive Training and Assess Neuroplasticity in Older Adults
Brief Title: Noninvasive Brain Stimulation to Enhance Cognitive Training in Older Adults
Acronym: MINDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 822954
Record Dates: First submitted 2019-07-30; First posted 2019-08-08 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Normal Aging
Keywords: non-invasive brain stimulation; cognition; transcranial direct current stimulation (tDCS)
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either receive real or sham tDCS without the option of crossover.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real tDCS + CBCT (Active Comparator): 20 minutes of 2.0mA of tDCS for 5 consecutive days
  Interventions: Device: Transcranial Direct Current Stimulation; Behavioral: Computer-based cognitive therapy (CBCT)
- Sham + CBCT (Sham Comparator): Sham stimulation closely imitates reals tDCS 30 second ramp-up / ramp-down
  Interventions: Device: Transcranial Direct Current Stimulation; Behavioral: Computer-based cognitive therapy (CBCT)

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — tDCS is a neuromodulatory technique that delivers a small electric current (about the equivalent of a 9V battery) to the head. A fixed current between 1 and 2 mA is typically applied. tDCS works by applying a positive (anodal) or negative (cathodal) current via electrodes to an area, facilitating the depolarization or hyperpolarization of neurons, respectively.
Behavioral: Computer-based cognitive therapy (CBCT) — Repetitive, drill-like training usually presented in the form of a game that targets a specific cognitive construct.

SUMMARY:
This research study explores the feasibility of pairing computer-based cognitive training (CBCT) with transcranial direct current stimulation (tDCS), a form of non-invasive brain stimulation, in order to enhance and preserve mental skills in older adults. The investigators aim to enhance participants ability to perform tasks of memory, attention, processing speed and other areas of cognition. Additionally, researchers are interested in the ability of the brain to adapt to change-neuroplasticity. Neuroplasticity is thought to impact how individuals respond to cognitive training and tDCS. In order to look at individual differences in neuroplasticity transcranial magnetic stimulation (TMS), a noninvasive brain stimulation technique, will be used. Individual responses to TMS can be used as a marker of neuroplastic changes in brain function, in order to reveal the relationship between brain plasticity and tDCS-induced changes in cognitive ability.

DETAILED DESCRIPTION:
Promising evidence suggests that cognitive training regimens may have some beneficial effects on cognition in older adults. However, the improvement from computer-based cognitive training (CBCT) diminish over time which highlights a fundamental challenge for CBCT interventions. Transcranial direct current stimulation (tDCS) can enhance certain cognitive skills, particularly when stimulation is combined with rehearsal of relevant behaviors. Importantly, these benefits have been shown to persist up to 2 months after the intervention.

This study will lay the groundwork for larger scale studies that will combine CBCT with neuromodulation, potentially leading to the development of a persistent, transferrable, multimodal technique to preserve cognition in older adults. In this study, participants will be randomly assigned to receive either real or sham tDCS for 5 consecutive days in conjunction with CBCT. The participant's cognition will be assessed with a neuropsychological assessment at baseline, 1 week, 2 weeks, and 2 months in order to determine any changes.

Additionally, transcranial magnetic stimulation (TMS) will be used to characterize the relationship between baseline differences in brain plasticity and cognitive changes induced by tDCS+CBCT. The effects of TMS on cortical activity have been shown to depend on a variety of neuroplasticity-related mechanisms. In this study, changes in motor physiology (called motor evoked potentials (MEPs)) induced by TMS will be used. Stimulation of the motor cortex with TMS induces robust, transient, and readily quantifiable changes in motor excitability, which are sensitive to changes in the mechanisms of neuroplasticity. Investigators hypothesize that individual variability in brain plasticity, measured by changes in MEP response to TMS, will predict the degree of cognitive benefit afforded by tDCS+CBCT.

Study Visits:

---------------- Visit 1 - Consent and Screening (2 hours) Review enrollment documents and conduct baseline neuropsychological assessment

---------------- Visit 2 - Visit 5 - tDCS + CBCT (30 minutes) Subjects will receive either real or sham stimulation along with cognitive training

--------------- Visit 6 - tDCS + CBCT & Follow-up (3 hours) Subjects will receive either real or sham stimulation along with cognitive training & follow-up neurospychological assessment

--------------- Visit 7 - TMS (3 hours) Subjects will receive TMS in order to induce MEPs

------------ Visit 8 - 2 week follow-up (1 .5 hours) Follow-up neuropsychological assessment

----------- Visit 9 - 2 month follow-up (1.5 hours) Follow-up neuropsycological assessment

ELIGIBILITY:
Inclusion Criteria:

* Normal cognition
* English as their native language

Exclusion Criteria:

1. . History of neurological disorders
2. . History of head injury with unconsciousness lasting more than 5 minutes
3. . History of psychiatric disorders
4. . Currently abusing alcohol or drugs (prescription or otherwise)
5. . History of epilepsy or seizures within the past 6 months
6. . Previous brain surgery
7. . Pacemaker

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-08-18 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Executive Function | baseline, day 5, 2 week, 2 months
  Change in tDCS induced executive function as measured by the Delis-Kaplan Executive Function Systems (DKEFS) test.
  DKEFS utilizes a scaled score which ranges from 1-20 with scores between 8-12 considered average.

SECONDARY OUTCOMES:
TMS brain activation | 2 week
  Change in average amplitude of MEPs as a response to TMS. We expect to see an initial reduction (or inhibition) in average amplitude of the MEP response to TMS, followed by a return to baseline amplitude.